CLINICAL TRIAL: NCT01319071
Title: Genetic Polymorphism and Israeli Top-level Athletes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Wingate Institute (Other)
Responsible Party: Eias Kassem, MD, Hillel Yaffe Medical Center
Other Study IDs: 0015-11-HYMC
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Top-level Athletes
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Top-level athletes
  Interventions: Other: Blood sample
- Control group
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Extraction of blood sample from top-level athletes

SUMMARY:
It is still unknown whether different genetic elements play a role in athletes' ability to create their area of specificity.In a study conducted in our laboratory few years ago, we genotyped 22 genes in 2 athletic groups (endurance and sprinters) and in age and gender matched nonathletic controls. Few of these genes were found to be associated with athletic performance and area of specificity. Since then a few more genes have been found that are related to athletic performance, and our aim in the current study is to expand our research to these new genes which include 3 genetic cascades: genes associated with body fluid balance and homeostasis, genes associated with muscle strength, and genes associated with bioenergy.

ELIGIBILITY:
Inclusion Criteria:

* Top-level athletes
* Other athletes

Exclusion Criteria:

* All others

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes training at the Wingate Institute
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genes related to top-level athletes | Four months

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate Institute, Netanya, Israel